CLINICAL TRIAL: NCT05226728
Title: Clinical Efficacy and Safety of Individual Pembrolizumab Administration Based on Pharmacokinetic in Advanced Non-small Cell Lung Cancer: an Open-label, Single Arm, Exploratory Clinical Trial
Brief Title: Pharmacokinetically-guided on the Individualization of Pembrolizumab Administration in the Treatment of Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO 1054
Record Dates: First submitted 2021-06-27; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Pembrolizumab; Pharmacokinetics; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pharmacokinetic-guided pembrolizumab cohort (Experimental): Eligible patients received pembrolizumab 200mg every 3 weeks with or without chemotherapy for four cycles, then for patients without progressive disease, pembrolizumab was administrated in new dose-intervals according to steady state plasma-concentration (Css) of pembrolizumab until disease progression.
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — Eligible patients received pembrolizumab 200mg every 3 weeks with or without chemotherapy for four cycles, then for patients without progressive disease, pembrolizumab was administrated in new dose-intervals according to steady state plasma-concentration (Css) of pembrolizumab until disease progression
  Other Names: keytruda

SUMMARY:
Pembrolizumab with or without chemotherapy has become the standard therapy in advanced non-small cell lung cancer (NSCLC), with a fixed dose of 200mg every 3 weeks. The investigators performed this study to explore the clinical efficacy and safety of pharmacokinetic (PK)-guided pembrolizumab administration in advanced NSCLC.

DETAILED DESCRIPTION:
In this prospective, open-label, single-arm exploratory study, the investigators enrolled advanced NSCLC patients without sensitizing EGFR or ALK mutation in Sun yat-sen university cancer center. Eligible patients received pembrolizumab 200mg every 3 weeks with or without chemotherapy for four cycles, then for patients without progressive disease, pembrolizumab was administrated in new dose-intervals according to steady state plasma-concentration (Css) of pembrolizumab until disease progression. Primary endpoint was the progression-free survival. Patients with Css of pembrolizumab also underthe investigatorsnt genetic polymorphism analysis of variable number of tandem repeats region (VNTR) in neonatal Fc receptor (FcRn).

ELIGIBILITY:
Inclusion Criteria:

1. cytologically or histologically confirmed primary NSCLC;
2. Stage IV primary NSCLC according to the International Association for the Study of Lung Cancer (IASLC) TNM Eighth Edition;
3. There must be at least one evaluable lesion judged according to RECIST1.1;
4. No sensitive mutation in EGFR and negative ALK rearrangement;
5. ≥18 years old;
6. The Eastern Cooperative Oncology Group (ECOG) physical status score was 0-2;
7. Life expectancy of more than 3 months;
8. Bone marrow and organs (liver and kidney) function well, which can meet the conventional conditions for chemotherapy: neutrophil count ≥1.5×109/ L, platelet count ≥75×109/ L, hemoglobin ≥9g/ dL, total bilirubin ≤1.5×ULN, transaminase ≤2.5×ULN, serum creatinine ≤1.5×ULN or creatinine clearance ≥45ml/min. (ULN: upper limit of normal value);
9. For female subjects of reproductive age, urine or serum pregnancy test should be negative within 7 days prior to receiving the first study drug administration (cycle 1, day 1).If a urine pregnancy test is not confirmed negative, a blood pregnancy test is required;For men, consent must be given to use appropriate methods of contraception or surgical sterilization during the trial and for 8 weeks after the last administration of the experimental drug;
10. Signing the informed consent;
11. Good compliance, follow-up, and voluntary compliance with relevant regulations of the study.-

Exclusion Criteria:

1. Small cell lung cancer;
2. Brain metastases with hemorrhage;
3. Currently participating in interventional clinical research and treatment;
4. Past anti-tumor immunotherapy with other anti-PD-1 /PD-L1 monoclonal antibodies;
5. Have received solid organ or blood system transplantation;
6. An active autoimmune disease requiring systemic treatment (e.g., use of palliative drugs, corticosteroids, or immunosuppressants) occurred within 2 years prior to initial administration.Alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic;
7. having been diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to the first administration of the study;Physiological dose of glucocorticoids (≤10 mg/ day of prednisone or its equivalent) is allowed;
8. A history of non-infectious pneumonia requiring glucocorticoid therapy or current interstitial lung disease within 1 year prior to initial administration;
9. A known history of human immunodeficiency virus (HIV 1/2 antibody positive);
10. untreated active hepatitis B

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
PFS | 18 months
  median progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Likun Chen, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang N, Zheng L, Li M, Hou X, Zhang B, Chen J, Li S, Chen L. Clinical efficacy and safety of individualized pembrolizumab administration based on pharmacokinetic in advanced non-small cell lung cancer: A prospective exploratory clinical trial. Lung Cancer. 2023 Apr;178:183-190. doi: 10.1016/j.lungcan.2023.02.009. Epub 2023 Feb 15. PMID 36868179